CLINICAL TRIAL: NCT04987619
Title: Acute Effects of Beetroot Juice Supplements on Lower-limb Strength and Muscular Endurance in Physically Active Women: Double-blind Crossover Randomized Trial
Brief Title: Effect of Beetroot Juice Supplements on Lower-limb Strength in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BEETROOT JUICE
Record Dates: First submitted 2021-07-20; First posted 2021-08-03 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-07

CONDITIONS: Muscular Endurance
Keywords: Explosive force production; Beetroot juice; Beetroot; muscular endurance

STUDY DESIGN:
Intervention Model Description: The experimental procedure will consist of three visits, separate from each other by one week, to achieve the total elimination of any effects caused by BJR as well as the optimal recovery of the participants.
Who Masked: Participant, Investigator
Masking Description: The order in which the participants will consume one supplement or another will be assigned randomly and double blind by an external collaborator to the research team, who will be responsible for coding the bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BJR (Experimental): 70 mL of beetroot juice (BEET It Sport®; James White Drinks Ltd., Ipswich, UK)
  Interventions: Dietary Supplement: Beetroot juice
- PLA (Placebo Comparator): 70 mL of blackcurrant beverage Capri-Sun.
  Interventions: Other: Capri-Sun

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Subjects will drink juice 120 minutes before each visit
  Arms: BJR
Other: Capri-Sun — 70 mL of blackcurrant beverage, which is depleted of NO3- will be taken 120 min before each visit.
  Arms: PLA

SUMMARY:
This study aims to evaluate the effects of beetroot juice supplements on lower-limb strength and muscular endurance in physically active women, due to the presence of NO3- in beetroot juice.

DETAILED DESCRIPTION:
Beetroot juice (BJR) is used as an ergogenic aid, but no study has analyzed its' effects on explosive force production in physically active women. It has been proposed that females could blunt reduction of NO2- to NO based on a higher oxidative skeletal muscle phenotype than males. However, it has been observed a higher increase on plasma NO2- levels after supplementation compared to and a greater enhancement on muscle contractile function.

Based on the absence of any study that has analyzed the effect of NO3- supplements on jump ability and power production on weightlifting on female population; the purpose of this study will be to investigate the possible ergogenic effect of BJR on physically active women on explosive force production and muscular endurance in a lower-limb body weightlifting protocol, due to the presence of NO3- in BJR and its effects.

ELIGIBILITY:
Inclusion Criteria:

* Physically active females with 18-30 years of age
* More than 6 months on RT training programs
* Be familiarized with back squat, leg press and leg extension exercises
* Not consuming any type of nutritional supplement or anabolic substances in the previous three months or during the study
* Not suffering from a musculoskeletal injury that could interfere with the exercise protocol during the investigation

Exclusion Criteria:

* None

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identity
Enrollment: 11 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Change of height reached in jump | Week 1, 2 and 3.
  Evaluated through CMJ (Counter movement jump) test with a recovery period of 45 seconds between jumps.

SECONDARY OUTCOMES:
Movement velocity | Visit 1 (week 1), 2 (week 2) and 3 (week 3).
  Evaluated at 50% and 75% repetition maximum (RM)
Power on back squat | Visit 1 (week 1), 2 (week 2) and 3 (week 3).
  Evaluated at 50% and 75% repetition maximum (RM)
Muscular endurance test | Visit 1 (week 1), 2 (week 2) and 3 (week 3).
  The test consists of three exercises: back squat, leg press and leg extension. Three series will be performed until concentric failure at 75% RM, three minutes of rest between each series.
Rating of perceived exertion (RPE). | Visit 1 (week 1), 2 (week 2) and 3 (week 3).
  Immediately at the end of the muscular endurance test, participants will be instructed to report their RPE using a scale 1-10 (worse to better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Jurado Castro, Principal Investigator — Hospital Universitario Reina Sofía
Locations (6):
- Studies Research Group in Neuromuscular Responses (GEPREN), University of Lavras, Lavras, Brazil
- Spain (5):
  - Maimonides Biomedical Research Institute of Cordoba (IMIBIC), Reina Sofia University Hospital, University of Cordoba, Córdoba
  - Metabolism and Investigation Unit, Maimonides Biomedical Research Institute of Cordoba (IMIBIC),Reina Sofia University Hospital, University of Cordoba, Córdoba
  - Department of Food Science and Technology, Rabanales University Campus, University of Cordoba, Córdoba
  - Department of Nursing Pharmacology and Physiotherapy, Faculty of Medicine and Nursing, University of Córdoba, Córdoba
  - Departamento de Motricidad Humana y Rendimiento Deportivo, Universidad de Sevilla, Seville

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the study concludes and results are published
Time Frame: After results are published
Access Criteria: Upon request to study's principal investigator